CLINICAL TRIAL: NCT02255214
Title: Evaluation of the Accuracy of the Hemochron Signature Elite Point of Care Micro Coagulation Instrument Compared With Laboratory Assay
Brief Title: Evaluation of the Accuracy of the Hemochron Signature Elite Point of Care Device Compared With Laboratory Assay
Status: Completed | Type: Observational
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2013/0300
Record Dates: First submitted 2014-02-14; First posted 2014-10-02 (Estimated); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Blood Coagulation Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical Patient: These are the results from the blood samples taken from the study participants.

SUMMARY:
Central Neuraxial Blockade (CNB) is commonly used in anaesthetics. It has several advantages over a general anaesthetic however contraindications include coagulopathy. Guidelines suggest a CNB should not be undertaken with an International Normalised Ratio (INR) of 1.5 or greater. A common cause of an elevated INR is warfarin therapy and regular monitoring of its effects is required.

The Hemochron Signature Elite is a portable micro coagulation system that can be used as a point of care (POC) anticoagulation monitoring device. Marketing is focussed on its accuracy, convenience and efficiency in delivering a coagulation result.

This study will assess the accuracy of this device in calculating the International Normalised Ratio (INR) result. This will be compared to another INR result obtained on the same sample via the current gold standard testing equipment in the Royal Infirmary Edinburgh (RIE) laboratories.

The study will include patients presenting for surgery who have had their warfarin therapy stopped within the previous 7 days. Patients on warfarin therapy requiring surgery are currently identified in preoperative assessment clinics, on average 12 weeks prior to their date of surgery.

Anecdotally there appears to be a difference between the 'expected' and actual INR when a POC device is used. Concern exists that patients may be inappropriately denied the potential benefits of central neural blockade (CNB) if a POC device provides a falsely high result, or conversely the investigators may be proceeding with CNB in patients with an unacceptably high INR if POC provides a falsely low result. There is also the possibility of improving hospital efficiency using this device as it provides a result much faster than the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting for elective surgery who have stopped their warfarin therapy within the last 7 days.

Exclusion Criteria:

* Adults with incapacity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all adult patients presenting for elective surgery who have stopped their warfarin therapy within the last 7 days. They will be approached in the Day Surgery Unit and Day of Surgery Assessment unit within a single centre.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cameron R Ferguson, MBChB MRCP, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, Lothian, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: The patients were collected as one group. Baseline characteristics were not obtained for this study as per the protocol. Each patient had one sample of blood taken, as per the study protocol. This blood sample was used for both the point of care coagulation testing device, and the laboratory coagulation test. No further intervention was taken place on any patient.
Period: Overall Study
Arm/Group | Group 1
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participant Group: Baseline characteristics for the participants were not recorded.
Arm/Group | Participant Group
Number analyzed (Participants) | 24
Age, Customized [Count of Participants; unit: Participants] — Population: Age data not collected
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/gender not recorded
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24

OUTCOME MEASURES:

1. Primary Outcome: The International Normalised Ratio (INR) Will be Measured by the Laboratory Assay and the Hemochron Signature Elite Device.
Description: The correlation between the international normalised ratio measured by the laboratory assay and the Hemochron Signature Elite device was assessed.Number of participants with a higher INR measurement by the Hemochron Signature Elite device than laboratory assay
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Primary Outcome Measure Results: All participants
Arm/Group | Primary Outcome Measure Results
Number analyzed (Participants) | 24
Participants | 23

ADVERSE EVENTS:
Groups:
- Adverse Events: There were no adverse events encountered.
Arm/Group | Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes